CLINICAL TRIAL: NCT07100730
Title: A Global, Multicenter, Prospective, Controlled, Open-Label Pivotal Study of Iodofalan (131I) Solution for Injection (TLX101-Tx) Plus Lomustine Versus Lomustine Alone in Patients With Radiographically Confirmed Recurrent Glioblastoma at First Recurrence (IPAX BrIGHT [IPAX-3])
Brief Title: Study of TLX101-Tx Plus Standard of Care (SoC) Versus SoC Alone for the Treatment of Patients With Recurrent Glioblastoma
Acronym: IPAX BrIGHT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 131I-TLX-101-003; 2025-521785-10 (EudraCT Number)
Record Dates: First submitted 2025-07-17; First posted 2025-08-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Neoplastic Disease; Glioblastoma; Glioblastoma (GBM); Glioblastoma Multiform; Glioblastoma Multiforme, Adult; Glioblastoma Multiforme (GBM) WHO Grade IV
Keywords: Lomustine; Radiation Therapy; Radiopharmaceuticals; Positron-Emission Tomography; Brain Neoplasms; Glioblastoma Multiforme; Glioblastoma; GBM; Neoplasm Recurrence, Local; Central Nervous System Neoplasms; Brain cancer; Recurrent brain tumor; Brain tumor recurrence; LAT-1 targeted therapy
MeSH Terms: conditions — Neoplasms; Glioblastoma; Brain Neoplasms; Neoplasm Recurrence, Local; Central Nervous System Neoplasms | interventions — Lomustine

STUDY DESIGN:
Intervention Model Description: In the first part of the trial, cohort of patients will receive different doses of the study drug and lomustine. If the drug is not well tolerated, the dose will change in new groups of patients and additional arms of the study will open. Doctors watch closely for any serious side effects, which helps them decide when the dose is too high.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLX101-Tx + Standard of Care (Experimental): TLX101-Tx + Lomustine
  Interventions: Combination Product: TLX-101-Tx + Lomustine
- TLX101-Tx Only (Experimental): TLX101-Tx Therapy only
  Interventions: Radiation: TLX101-Tx

INTERVENTIONS:
Combination Product: TLX-101-Tx + Lomustine — Combination therapy with TLX-101-Tx + Lomustine
  Other Names: 131I-IPA; 131I-TLX101
  Arms: TLX101-Tx + Standard of Care
Radiation: TLX101-Tx — TLX101-Tx
  Other Names: 131I-IPA; 131I-TLX101
  Arms: TLX101-Tx Only

SUMMARY:
This global clinical trial which evaluates the efficacy and safety of TLX101-Tx, an investigational radiopharmaceutical therapy, in combination with lomustine versus lomustine alone in adult patients with first recurrence of glioblastoma. TLX101-Tx delivers targeted radiation to glioblastoma cells. The trial is conducted in two parts: Part 1 assesses safety and radiation dosing; Part 2 is a randomized comparison of the combination therapy against standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Previously confirmed neuropathological diagnosis of glioblastoma, IDH-wildtype according to the WHO 2021 classification.
2. Radiographic evidence of first recurrence or progressive glioblastoma according to RANO 2.0 criteria after first-line treatment with biopsy or maximal safe resection and standard radiotherapy or chemoradiotherapy having occurred at least 3 months after the end of prior radiotherapy. Prior first-line therapy may include a combination of:

   1. Any systemic antineoplastic treatment other than nitroureas
   2. Tumor-treating fields
   3. Conventionally fractionated or abbreviated (minimum 15 fractions) radiotherapy
3. Increased [18F]]FET PET tracer uptake inside or in the vicinity of tumor. Specifically, amino acid-based molecular imaging using [18F]FET PET will be evaluated following co-registration with MRI. The allocated physician/reader will assess whether the observed pathologically increased amino acid uptake is located within the tumor or in the vicinity. This determination will serve as a guidance to confirm whether the uptake is tumor-associated. The uptake must be clearly discernible from background activity and measurable per PET RANO 1.0 criteria, as determined by central review.
4. Tumor debulking for recurrent, progressive disease is allowed. The patient must have post-surgical (4-6 weeks) radiographic evidence for residual tumor according to RANO 2.0 with increased [18F] FET PET uptake and measurable disease according to PET RANO 1.0.
5. 18 years or older
6. Have the capacity to understand the study and be willing to comply with all protocol requirements.
7. Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2 or KPS≥70
8. Patients on stable, not increasing dose of steroids in the previous 7 days can be included in the study
9. Adequate hematological, liver and renal function at the time of screening.
10. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of investigational drug product; must not be breast-feeding; and must agree to use a highly effective method of contraception during treatment and for 6 months following last dose of investigational product.
11. Male patients must agree to use condoms during sex during the treatment period and for 3 months after the last dose of the investigational drug product and must not make semen donations during treatment and for 6 months following last dose of investigational drug product. For male patients with female partners of childbearing potential, females must agree to use a highly effective method of contraception during the treatment period and for 6 months following last dose of investigational drug product.

Exclusion Criteria:

1. Prior course with external beam radiation to the brain in the past 3 months. Prior treatment with brachytherapy in the brain.
2. Treatment with bevacizumab within the prior 6 weeks.
3. Known contraindication to imaging tracer or any product of contrast media and MRI contraindications including implanted medical devices. Unable to lie still for at least 20 min or the duration of the MRI and PET imaging or the need for general anesthesia as part of the imaging procedure.
4. History or evidence of delayed-type hypersensitivity-dependent chronic infection (ie, tuberculosis, systemic fungal or parasitic infection).
5. Radiographic progression based on RANO 2.0 associated with clinical deterioration and life expectancy less than 3 months.
6. Hemostaseologic conditions, precluding catheterization or invasive procedures.
7. Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product.
8. Known liver or kidney disease, such as hepatitis, cirrhosis, renal failure.
9. Severe chronic or active infections (including active tuberculosis, hepatitis B virus, or hepatitis C virus infection) requiring systemic therapy.
10. Ongoing toxicity > Grade 2 NCI-CTCAE (version 5.0) from previous standard or investigational therapies.
11. Administration of another investigational product within 90 days prior to screening.
12. Expected non-compliance with longer-term admission at isolated nuclear medicine ward per regional regulations.
13. Inability to complete the needed investigational and standard imaging examinations due to any reason (ie, severe claustrophobia, inability to lie still for the entire imaging time).
14. Patients with known phenylketonuria.
15. Presence of any other condition that may increase the risk associated with study participation or interfere with the interpretation of study results, and, in the opinion of the study investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, an average of 2 years
  Assessing TEAEs type according to MedDRA (Medical Dictionary for Regulatory Activities), frequency, severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V5.0, seriousness, and relationship of study treatment will be assessed. Laboratory abnormalities will be assessed according to the NCI CTCAE V5.0.
Dose Optimization | Through study completion, an average of 2 years
  Part 1 of the study is being done to identify the best dose to use for Part 2 of the study

SECONDARY OUTCOMES:
TLX101-Tx Concentration in the blood | From enrollment to the end of treatment at around 12 weeks.
  Monitor how TLX101-Tx and its radioactive component move through the body over time. This includes checking how much of it is found in the blood at different times.
Radiation Dosimetry | Through study completion, an average of 2 years
  We will measure how much radiation from TLX101-Tx reaches the tumor and the bone marrow. This is done using special imaging scans (called SPECT, CT, and MRI) that help us see where the treatment goes in the body.
TLX101-Tx Concentration in the Urine | From enrollment to the end of treatment at around 12 weeks.
  Monitor how TLX101-Tx and its radioactive component move through the body over time. This includes checking how much is passed out in urine at different times following treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Austin Health, Melbourne
  - Royal North Shore Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No
We have opted not to share individual participant data due to concerns regarding participant privacy and the absence of explicit consent for data sharing in the original trial protocol especially for patients enrolled in the EU.